CLINICAL TRIAL: NCT05055258
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial to Evaluate the Efficacy and Safety of 3 Dose Levels of KVD824, an Oral Plasma Kallikrein Inhibitor, for Long-Term Prophylactic Treatment of Hereditary Angioedema Type I or II
Brief Title: A Trial to Evaluate the Efficacy and Safety of Different Doses of KVD824 for Prophylactic Treatment of HAE Type I or II
Acronym: KVD824-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor due to adverse events reported
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KVD824-201
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Angioedema, Hereditary, Types I and II
Keywords: KVD824; KOMPLETE
MeSH Terms: conditions — Hereditary Angioedema Types I and II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 300 mg KVD824 (Experimental): 300 mg KVD824 twice a day for 12 weeks
  Interventions: Drug: KVD824
- 600 mg KVD824 (Experimental): Two 300 mg KVD824 tablets twice a day for 12 weeks
  Interventions: Drug: KVD824
- 900 mg KVD824 (Experimental): Three 300 mg KVD824 tablets twice a day for 12 weeks
  Interventions: Drug: KVD824
- Placebo to KVD824 (Placebo Comparator): One, two or three placebo tablets to be taken twice a day for 12 weeks
  Interventions: Drug: Placebo to KVD824

INTERVENTIONS:
Drug: KVD824 — KVD824 300 mg Modified-Release Tablets
  Arms: 300 mg KVD824; 600 mg KVD824; 900 mg KVD824
Drug: Placebo to KVD824 — Placebo to KVD824 300 mg Modified-Release Tablets
  Arms: Placebo to KVD824

SUMMARY:
A study to assess whether different doses of KVD824 are effective in preventing attacks of Hereditary Angiodedema Type I or Type II.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age and older.
2. Confirmed diagnosis of HAE type I or II at any time in the medical history:

   1. Documented clinical history consistent with HAE (subcutaneous or mucosal, nonpruritic swelling episodes without accompanying urticaria) AND EITHER
   2. Diagnostic testing results obtained prior to randomization that confirm HAE Type I or II: C1-INH functional level <40% of the normal level. Subjects with functional C1-INH level 40-50% of the normal level may be enrolled if they also have a C4 level below the normal range. Testing may be obtained from central or local laboratories or obtained from documented historical testing results. Subjects may be restested at anytime prior to randomization if results are incongruent with clinical history or believed by the Investigator to be confounded by recent prophylactic or therapeutic C1 INH use, OR
   3. Documented genetic results that confirm known mutations for HAE Type I or II.
3. Subject has access to and ability to use conventional treatment for HAE attacks.
4. Subject is willing to cease any current medications being taken for HAE prophylaxis and Investigator determines that doing so would not place the subject at any undue safety risk.
5. Subject's last dose of attenuated androgens was at least 28 days prior to first dose of IMP.
6. During the Run-in Period subject meets one of the following criteria:

   1. Two Investigator-confirmed attacks in the first 4-week period.
   2. Three Investigator-confirmed attacks in ≤8 weeks.
7. Subjects who are fertile and heterosexually active must adhere to contraception requirements throughout the trial as follows:

   a) Female subjects must agree to use at least one highly effective contraception method from the Screening Visit until the end of the trial. Highly effective methods of contraception include: i) Progestogen-only hormonal contraception associated with inhibition of ovulation: oral/injectable/implantable (hormonal contraception that contains estrogen including ethinylestradiol is excluded per Exclusion 4).

   ii) Intrauterine device (IUD). iii) Intrauterine hormone-releasing system (IUS). iv) Bilateral tubal occlusion. v) Vasectomized partner (provided that the partner is the sole sexual partner of the female subject of childbearing potential and that the vasectomized partner has received medical assessment of surgical success).

   b) Male subjects with a female partner of childbearing potential must agree to use condoms for the entire Treatment Period AND for 90 days following the final dose of investigational medicinal product (IMP). Female partners are encouraged to use contraception as outlined in Inclusion 7a) from the Screening Visit until the end of the trial. Hormonal contraception that contains estrogen including ethinylestradiol is acceptable for the female partner.
8. Subjects who are not fertile or not sexually active, as defined below, do not require contraception.

   1. Subjects who refrain from heterosexual intercourse during the trial if the reliability of the heterosexual abstinence has been evaluated in relation to the duration of the clinical trial and is the preferred and usual lifestyle of the subject.
   2. Male subjects who are surgically sterile (e.g. vasectomized with medical assessment of surgical success).
   3. Female subjects who are surgically sterile (e.g. status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post menopausal for at least 12 months.
9. Subjects must be able to swallow trial tablets whole.
10. Subjects assessed by the Investigator must be able to appropriately receive and store IMP, and be able to read, understand, and complete the eDiary.
11. Investigator believes that the subject is willing and able to adhere to all protocol requirements.
12. Subject provides signed informed consent and is willing and capable of complying with trial requirements and procedures.

Exclusion Criteria

1. Any concomitant diagnosis of another form of chronic angioedema, such as acquired C1 inhibitor deficiency, HAE with normal C1-INH (previously known as HAE type III), idiopathic angioedema, or angioedema associated with urticaria.
2. A clinically significant history of poor response to C1-INH therapy or plasma kallikrein inhibitor therapy for the management of HAE, in the opinion of the Investigator.
3. Use of angiotensin converting enzyme (ACE) inhibitors after the Screening Visit or within 7 days prior to randomization.
4. Any estrogen containing medications with systemic absorption (such as oral contraceptives including ethinylestradiol or hormonal replacement therapy) after the Screening Visit or within 7 days prior to randomization.
5. Use of narrow therapeutic index drugs metabolized by CYP3A4 or CYP2C9 or transported by OAT1, OCT2, and OATP1B1, starting at screening, as determined by the Investigator.
6. Use of strong CYP3A4 inhibitors and inducers during participation in the trial, starting at the Screening Visit.

   Note: These medications include but are not limited to the following:

   Inhibitors: boceprevir, clarithromycin, cobicistat, dasabuvir, denoprevir, elvitegravir, idelalisib, indinavir, itraconazole, ketoconazole, lopinavir, nefazodone, nelfinavir ombitasvir, paritaprevir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, tipranavir, troleandomycin, and voriconazole.

   Inducers: apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's Wort.
7. Inadequate organ function, including but not limited to;

   1. Alanine aminotransferase (ALT) > 2x Upper limit of Normal (ULN).
   2. Aspartate aminotransferase (AST) > 2x ULN.
   3. Bilirubin direct > 1.25x ULN.
   4. International normalized ratio (INR) > 1.2.
   5. Clinically significant hepatic impairment defined as a Child-Pugh B or C.
   6. Estimated glomerular filtration rate (eGFR) <60 mL/min.
8. Any clinically significant comorbidity or systemic dysfunction that in the opinion of the Investigator would jeopardize the safety of the subject by participating in the trial.
9. History of substance abuse or dependence that would interfere with the completion of the trial, as determined by the Investigator.
10. Known hypersensitivity to KVD824 or placebo or to any of the excipients.
11. Any prior use of any gene therapy treatment for HAE.
12. Participation in any interventional investigational clinical trial, including an investigational COVID-19 vaccine trial, within 4 weeks of the last dosing of investigational drug prior to screening.
13. Any pregnant or breastfeeding subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
The Rate of Investigator-confirmed HAE attacks during the Treatment Period | 12 weeks
  To examine the number of investigator-confirmed attacks whilst on treatment compared to placebo

SECONDARY OUTCOMES:
Proportion of subjects without Investigator-confirmed HAE attacks during the Treatment Period. | 12 weeks
Rate of Investigator-confirmed HAE attacks that require conventional treatment during the Treatment Period. | 12 weeks
Angioedema Quality of Life Questionnaire (AE-QoL) total score and domain scores during the Treatment Period. | 12 weeks
  AE-QoL is a quality of life questionnaire with a range of 0 (minimum) to 100 (maximum). A total score of 100 indicates worst possible impairment.
Angioedema Control Test (AECT) score and domain scores during the Treatment Period. | 12 weeks
  AECT is a 4-item patient-reported outcome measure. The total score is from 0 (minimum) to 16 (maximum). A higher score indicates a higher level of angioedema control.
Proportion of subjects with an AECT score ≥12 at the end of the Treatment Period. | 12 weeks
  AECT is a 4-item patient-reported outcome measure. The total score is from 0 (minimum) to 16 (maximum). A higher score indicates a higher level of angioedema control.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals
Locations (33):
- United States (13):
  - KalVista Investigative Site, Birmingham, Alabama
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, La Jolla, California
  - KalVista Investigative Site, Santa Monica, California
  - KalVista Investigative Site, Centennial, Colorado
  - KalVista Investigative Site, Tampa, Florida
  - KalVista Investigative Site, Chevy Chase, Maryland
  - KalVista Investigative Site, Boston, Massachusetts
  - KalVista Investigative Site, St Louis, Missouri
  - KalVista Investigative Site, Cincinnati, Ohio
  - KalVista Investigative Site, Hershey, Pennsylvania
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investigative Site, Spokane, Washington
- KalVista Investigative Site, Campbelltown, New South Wales, Australia
- KalVista Investigative Site, Sofia, Bulgaria
- KalVista Investigative Site, North York, Ontario, Canada
- Czechia (2):
  - KalVista Investigative Site, Brno
  - KalVista Investigative Site, Prague
- France (2):
  - KalVista Investigative Site, Grenoble
  - KalVista Investigative Site, Paris
- Germany (3):
  - KalVista Investigative Site, Mainz, Rhineland-Palatinate
  - KalVista Investigative Site, Berlin
  - KalVista Investigative Site, Frankfurt am Main
- KalVista Investigative Site, Budapest, Hungary
- Italy (2):
  - KalVista Investigative Site, Milan
  - KalVista Investigative Site, Padua
- KalVista Investigative Site, Grafton, Auckland, New Zealand
- KalVista Investigative Site, Skopje, North Macedonia
- KalVista Investigative Site, San Juan, Puerto Rico
- United Kingdom (4):
  - KalVista Investigative Site, Birmingham
  - KalVista Investigative Site, Leeds
  - KalVista Investigative Site, London
  - KalVista Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT05055258/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05055258/SAP_001.pdf